CLINICAL TRIAL: NCT06038643
Title: The Healthy Aging Brain Study: A Remote Behavioral Intervention to Enhance Physical Activity in Older Adults.
Brief Title: Intergenerational Behavioral Intervention to Enhance Physical Activity in Older Adults at Risk for Alzheimer's Disease
Acronym: HABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Montreal Neurological Institute and Hospital (Other); McGill University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maiya R. Geddes, MD, Assistant Professor, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUSMD-20-38; P30AG048785 (NIH)
Record Dates: First submitted 2022-04-25; First posted 2023-09-15 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Physical Inactivity
Keywords: Risk Factors; Disease Prevention; Alzheimer's Disease; Motivation
MeSH Terms: conditions — Sedentary Behavior; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Intergenerational Social Motivation Behavioral Intervention using a Technology-based Platform
  Our research will test an innovative, technology-based, and readily scalable cross-generational social behavior intervention to enhance physical activity in at-risk older adults through a randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Social motivation intervention, self-transcendence daily messages, and daily accelerometry.
  Interventions: Behavioral: Motivational behavioural intervention and daily activities monitoring
- Active Control (Active Comparator): Daily accelerometry.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Motivational behavioural intervention and daily activities monitoring — Social motivation manipulation, self-transcendence daily messaging, and daily activities monitoring through accelerometry. Participants in this arm will have a study partner who receives daily feedback on the main participant's daily step count.
  Arms: Intervention
Behavioral: Active Control — Daily activities monitored through accelerometry.
  Arms: Active Control

SUMMARY:
This is a four-week pilot randomized controlled trial of a behavioral intervention in older adults at risk for Alzheimer's disease. Older participants are a subgroup from the PREVENT-AD longitudinal cohort. We will test whether a four-week intergenerational social motivation using a technology-based platform (intervention group) enhances physical activity relative to a control group.

DETAILED DESCRIPTION:
This study is a two-arm, single-site randomized controlled trial to test whether a four-week technology-based intergenerational social motivation intervention enhances physical activity in 60 cognitively unimpaired older adults with a first-degree history of Alzheimer's disease. These at-risk older adults will be recruited as a subgroup from a longitudinal cohort at McGill University, PREVENT-AD. At the outset, half of the participants will be randomized to the intergenerational social motivation condition (intervention group) and the other half will be randomized to the control group (1:1). A multimodal AD risk score based on older participants' already acquired AD biomarker, health and cognitive data will be used as strata for randomization to ensure equal assignment of high-risk participants to Intervention and control groups, using a permuted block method with random blocks.

The primary outcome is an increase in step count as measured by accelerometer. Secondary outcomes are an increase in total physical activity, mood, generativity, cognition, and loneliness. After an initial visit consisting of behavioral testing and structural and functional MRI, participants in the intervention group will be paired with younger adults (14 to 40 years) to form intergenerational dyads. Younger adults are either a family member of the older adult or a younger adult recruited from the community. Participants in the intervention group will receive personalized, positive daily messages over a four-week period via their device using the 'Our Family Garden' technology platform. These daily messages combine (1) pro-social goals (donation to charity after reaching exercise goals), (2) intergenerational social engagement, and (3) positive personalized messages from their younger study partners. This study will have 6 visits over a 2-month period in addition to the four-week intervention period (3 months total). Cognitive and behavioral data will be collected at each visit and physical activity data will be collected over the intervention period.

The primary endpoint is defined as the end of the initial period. Data collected are stored in one of three ways; (1) Physical activity monitoring data are extracted from their respective software packages and uploaded directly to a secure data storage environment at a high-performance computing facility. All pen-and-paper psychosocial and neuropsychological assessments are scored and entered in REDCap. Computerized psychosocial assessments are collected directly in REDCap and computerized neuropsychological assessments are entered in REDCap. TextMagic is used to distribute the daily intervention messages. Collected and anonymized survey data are stored on the web application behind an administrative login developed with Django, a high-level Python web framework. All data from REDCap will be exported to CSV files using the data de-identification feature for subsequent analysis with R and SPSS statistical analysis packages. After compiling all data across the 3 different data servers, data will be checked for completeness and correctness using frequency distributions (for missing data and out-of-range values). For the final dataset, the multiple imputations by chained equations (MICE) will be used to input missing values with 10 imputations.

ELIGIBILITY:
Main Participant Inclusion criteria:

Men and women > 60 years Who are current participants of the PREVENT-AD Longitudinal Cohort at McGill University.

No contraindications to MRI Imaging. Normal cognition Not exercising more than 150 minutes of moderate-intensity exercise per week or sitting more than 8 hours per day AND responded "yes" to the question "Do you want to increase your physical activity?" Fluency in English or French Access to a computer or smartphone with internet Normal or corrected-to-normal vision based on the minimal 20/20 standard Ambulatory without significant increase in pain with walking or the assistance of walking devices

Main Participant Exclusion Criteria:

Primary care physician does not approve additional physical activity An inability to ambulate without the assistance of another person or severe pain

Any unstable medical condition:

* History of a psychiatric illness including schizophrenia or Attention Deficit Hyperactivity Disorder (ADHD). History of anxiety or depression accepted if stable on medication for at least 6 months
* Current treatment for cancer - except non-melanoma skin cancer
* Neurological condition (e.g., multiple sclerosis, Parkinson's disease, and stroke)
* Current alcohol or substance abuse
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, Deep Venous Thrombosis (DVT) or other unstable cardiovascular condition
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac event in the past six months.

Younger Adult Inclusion Criteria:

* Can be identified as child or grandchild of participant (biological or adopted), 14 years or older.
* Can be a young adult (18 years or older) who is not a relative of the main participant, in case a grandchild or child is not available.
* Stable on antidepressants for more than 6 months.
* In contact with the primary participant more than once per 12 months at baseline
* Lives anywhere in Canada if 18 years and older, or anywhere accessible by mail in Quebec if 14 years and older but younger than 18 years.
* Normal or corrected-to-normal vision based on the minimal 20/20 standard to complete the cognitive tasks
* Able to speak, read, and write English or French
* No diagnosis of neurological disease or unstable health condition

Study Partner Exclusion Criteria:

• Not in contact with the primary participant more than once per 12 months at baseline

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maiya R Geddes, MD PhD, Principal Investigator — McGill University
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Active Control
Started | 36 | 40
Completed | 26 | 36
Not Completed | 10 | 4
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Excluded (not longer fulfilled enrollment criteria) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Active Control | Total
Number analyzed (Participants) | 26 | 36 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 22 | 32 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.81 (4.32) | 70.97 (5.36) | 70.48 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 29 | 44
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 36 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 36 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 36 | 62
Years of Education [Mean (Standard Deviation); unit: years] | 16.08 (3.07) | 15.97 (3.55) | 16.02 (3.33)
APOE4 genotype [Count of Participants; unit: Participants] — The APOE gene provides instructions for making a protein that carries cholesterol in the blood. People inherit two copies of this gene, one from each parent, and there are different versions (called alleles): ε2, ε3, and ε4. The combination of these alleles is called a person's APOE genotype (for example, ε3/ε4). This genetic information can influence a person's risk of developing conditions like Alzheimer's disease.
  Collection Method: A blood sample is collected at the beginning of the study. DNA is extracted and tested in a laboratory to determine which APOE alleles a person has.
  Participants
    APOE4 carriers | 8 | 16 | 24
    APOE4 non-carriers | 18 | 20 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 27.39 (5.03) | 26.48 (4.56) | 26.86 (4.74)
Alzheimer's Disease Risk [Count of Participants; unit: Participants]
  Lower Risk | 18 | 19 | 37
  Higher Risk | 8 | 17 | 25
Mild Cognitive Impairment [Count of Participants; unit: Participants]
  Mild Cognitive Impairment | 6 | 6 | 12
  Cognitively Unimpaired | 20 | 30 | 50
Language [Count of Participants; unit: Participants]
  English | 4 | 5 | 9
  French | 22 | 31 | 53
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.69 (8.14) | 74.42 (6.58) | 74.53 (7.21)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125.81 (16.36) | 128.22 (14.79) | 127.21 (15.38)
Steps per day [Mean (Standard Deviation); unit: Steps/day] — "Steps per day" was defined as the mean number of steps across a minimum of 4 valid days within a 7-day period, based on daily accelerometry data.
  Steps/day | 4224.77 (3149.72) | 3881.07 (2978.81) | 4025.20 (3051.94)
TMB Serial Reaction Time [Mean (Standard Deviation); unit: seconds] — The TMB Serial Reaction Time task measures implicit sequence learning and visuomotor speed by tracking how quickly participants respond to repeating versus random visual cues.
  In the TMB Serial Reaction Time task, higher scores in seconds (i.e., longer reaction times) indicate:
  * Reduced processing speed
  * Lower motor or attentional efficiency
  * Weaker implicit sequence learning
  seconds | 364.73 (74.73) | 388.13 (103.15) | 378.54 (92.6)
TMB Choice Reaction Time [Mean (Standard Deviation); unit: seconds] | 1208.83 (327.14) | 1304.72 (639.63) | 1265.42 (532.66)
Test my Brain Gradual Onset Continuous Performance Test (C) [Mean (Standard Deviation); unit: Score on a scale] — This cognitive test battery contains Test my Brain (TMB) Gradual Onset Continuous Performance Test. In this go/no-go test, the participant presses a button for each city image and withholds button presses for mountain images. This is a test of cognitive control, sustained attention, and response inhibition. Values can be from -1.5 to +1.5. Higher scores indicate better performance. The CPT.C score is a measure of response criterion, or how quickly and/or impulsively the participant tended to respond. Higher scores represent greater response impulsivity.
  Score on a scale | 0.38 (0.43) | 0.33 (0.43) | 0.35 (0.43)
TMB Gradual Onset Continuous Performance Test (D) [Mean (Standard Deviation); unit: scores on a scale] — This cognitive test battery contains Test my Brain (TMB) Gradual Onset Continuous Performance Test. In this go/no-go test, the participant presses a button for each city image and withholds button presses for mountain images. This is a test of cognitive control, sustained attention, and response inhibition. The CPT.D score is a measure of discrimination performance, related to how accurately the participant was able to respond to mountains and scenes. Higher scores represent better performance. Values can be from 1 to 4. Higher scores indicate better performance.
  scores on a scale | 2.71 (0.77) | 2.58 (0.96) | 2.64 (0.88)
Test my Brain Matrix Reasoning [Mean (Standard Deviation); unit: Score on a scale] — In TMB Matrix Reasoning, the participant selects which smaller image completes the pattern in the larger image. This is a test of visual reasoning and general cognitive ability. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 2 to 32. Higher scores are better.
  Score on a scale | 21.4 (7.8) | 21.14 (6.8) | 21.25 (7.17)
Test my Brain Forward Digit Span [Mean (Standard Deviation); unit: Score on a scale] — In the forward version of TMB Digit Span, the participant is shown a series of numbers in increasing length and asked to recall the numbers in the order displayed. This is a test of short-term memory. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 1 to 11. Higher scores are better.
  Score on a scale | 6.84 (1.57) | 6.0 (1.99) | 6.35 (1.86)
Test my Brain Backwards Digit Span [Mean (Standard Deviation); unit: Score on a scale] — In the backward version, the participant is shown a series of numbers in increasing length and asked to recall the numbers in reverse order. This is a test of short-term memory and working memory. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 1 to 10. Higher scores are better.
  Score on a scale | 5.28 (1.88) | 4.94 (1.76) | 5.08 (1.81)
Test my Brain Visual Paired Associates Matching [Mean (Standard Deviation); unit: Score on a scale] — This cognitive testing battery contains Test my Brain (TMB) Visual Paired Associates Memory. In this test, the participant memorizes a set of picture pairs. Then, after completing TMB Digit Symbol Matching (90 sec), the participant selects which pictures were paired together. TMB Visual PA is a test of visual episodic memory. In TMB Digit SM, the participant matches as many number/symbol pairs as possible in 90 seconds. This is a test of processing speed. Scores go from 4 to 23. Higher scores are better.
  Score on a scale | 14.5 (4.3) | 14.9 (4.3) | 14.73 (4.3)
Test my Brain Digit Symbol Matching [Mean (Standard Deviation); unit: Score on a scale] — In TMB Digit Symbol Matching, the participant matches as many number/symbol pairs as possible in 90 seconds. This is a test of processing speed. This test was adapted from the Wechsler Adult Intelligence Scales. Higher scores are better. Scores go from 11 to 55.
  Score on a scale | 36 (6.95) | 35.53 (8.85) | 35.72 (8.06)

OUTCOME MEASURES:

1. Primary Outcome: Total Step Count (Average Steps/Day)
Description: This metric quantifies the change in the average number of steps taken each day, from the baseline period to the 4-week period. It is a marker of change in habitual ambulatory activity.
Time Frame: 4-week
Population: Participants included in the analysis were those who completed the study.
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 26 | 36
Steps/day | 5648.91 (4033.49) | 3809.62 (2833.25)
Statistical Analysis 1: Comparison: Intervention vs Active Control; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — Adjusted for multiple comparisons using False Discovery Rate

2. Secondary Outcome: The Modified Differential Emotions Scale (mDES) Negative Emotions
Description: The Modified Differential Emotions Scale (mDES) Negative Emotions subscale measures the intensity of negative emotional experiences such as sadness, anger, fear, and shame.
  Possible scores: min. 0, max. 80 A higher score indicates greater emotional intensity or frequency of the emotions assessed.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 23 | 31
score | 1.18 (0.27) | 1.31 (0.37)

3. Secondary Outcome: Generativity - Achievement
Description: This questionnaire measures generativity, which refers to the concern or desire individuals have to contribute to the well-being and development of future generations.
  Generative evaluates the extent to which individuals are motivated by generative concerns, including the desire to impact others and future generations; the Achievement subscale specifically captures the orientation toward personal goal attainment, mastery, and the pursuit of success as expressions of generativity.
  Scores for the generative achievement subscale ranged between 6 and 36, with higher scores indicating greater generative achievement.
Time Frame: 4 weeks
Population: Participants included in the analysis were those who completed the Generativity questionnaire.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
score | 25.09 (5.18) | 22.58 (5.88)

4. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Backwards Digit Span
Description: The TestMyBrain Digital Neuropsychology Toolkit Backwards Digit Span assesses working memory by requiring individuals to recall sequences of numbers in reverse order.
  In the backward version, the participant is shown a series of numbers in increasing length and asked to recall the numbers in reverse order. This is a test of short-term memory and working memory. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 1 to 10. Higher scores are better.
Time Frame: 4 weeks
Population: The population included in the analysis were those who completed the Test My Brain Backward Digit Span subtest.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 24 | 28
score | 6.58 (1.53) | 4.89 (1.83)
Statistical Analysis 1: Comparison: Intervention vs Active Control; We conducted one-way analyses of covariance (ANCOVAs) to assess the effect of group (intervention vs. control) on post-intervention secondary outcomes, including cognition (Test My Brain Digital Neuropsychology Toolkit). Covariates in all models included age, sex, years of education, APOE4 status, and baseline scores; Test type: Superiority; p < 0.01, ANCOVA

5. Secondary Outcome: Loneliness
Description: University of California, Los Angeles (UCLA) Loneliness Scale. A higher average score indicates greater loneliness. Possible scores: min. 20, max. 80.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 26 | 36
score | 53.71 (23.89) | 44.87 (19.25)

6. Secondary Outcome: Modified Differential Emotions Scale (mDES) Positive Emotions
Description: The Modified Differential Emotions Scale (mDES) Positive Emotions subscale measures the intensity of positive emotional experiences such as joy, gratitude, love, and hope.
  Possible scores: min. 0, max. 80 A higher score indicates greater emotional intensity or frequency of the emotions assessed.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 23 | 31
score | 3.38 (0.69) | 3.40 (0.75)

7. Secondary Outcome: Generativity Desire
Description: The Generative Test measures generativity, which refers to the concern or desire individuals have to contribute to the well-being and development of future generations. The Desire subscale specifically assesses the emotional motivation and intrinsic longing to nurture, support, and positively impact others and future generations.
  Scores for the generative desire subscale ranged between 7 and 42, with higher scores indicating greater generative desire.
Time Frame: 4 weeks
Population: Participants included in the analysis had completed the Generativity questionnaire.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
score | 31.67 (6.13) | 29.72 (7.05)

8. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Choice Reaction Time
Description: The TestMyBrain Digital Neuropsychology Toolkit Choice Reaction Time task measures processing speed and attention by assessing how quickly individuals respond to different stimuli.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Test My Brain Choice Reaction Time.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
seconds | 1293.08 (722.89) | 1136.67 (389.61)

9. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Digit Symbol Matching
Description: The TestMyBrain Digital Neuropsychology Toolkit Digit Symbol Matching task measures processing speed, attention, and visual-motor coordination by requiring rapid matching of symbols to corresponding numbers.
Time Frame: 4 weeks
Population: Participants included in the analysis had completed the Test My Brain Digit Symbol Matching subtest.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 20 | 28
score | 38.81 (7.14) | 36.83 (7.85)

10. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Forward Digit Span
Description: The TestMyBrain Digital Neuropsychology Toolkit Forward Digit Span task measures short-term memory by requiring individuals to recall sequences of numbers in the order presented.
  In the forward version of TMB Digit Span, the participant is shown a series of numbers in increasing length and asked to recall the numbers in the order displayed. This is a test of short-term memory. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 1 to 11. Higher scores are better.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Forward Digit Span.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 28
score | 6.91 (1.57) | 6.18 (1.81)

11. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Gradual Onset Continuous Performance C
Description: The TestMyBrain Digital Neuropsychology Toolkit Gradual Onset Continuous Performance Task measures sustained attention and inhibitory control by requiring individuals to detect target stimuli amid gradually changing non-targets.
  In this go/no-go test, the participant presses a button for each city image and withholds button presses for mountain images. This is a test of cognitive control, sustained attention, and response inhibition. Values can be from -1.5 to +1.5. Higher scores indicate better performance. The CPT.C score is a measure of response criterion, or how quickly and/or impulsively the participant tended to respond. Higher scores represent greater response impulsivity.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Test My Brain Gradual Onset Continuous Performance C subtest.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
score | 0.45 (0.25) | 0.40 (0.36)

12. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Gradual Onset Continuous Performance D
Description: The TestMyBrain Digital Neuropsychology Toolkit Gradual Onset Continuous Performance Task (D) assesses sustained attention and response inhibition by requiring individuals to monitor and respond to target stimuli within a dynamic visual stream.
  In this go/no-go test, the participant presses a button for each city image and withholds button presses for mountain images. This is a test of cognitive control, sustained attention, and response inhibition. The CPT.D score is a measure of discrimination performance, related to how accurately the participant was able to respond to mountains and scenes. Higher scores represent better performance. Values can be from 1 to 4. Higher scores indicate better performance.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Test My Brain Gradual Onset Continuous Performance D subtest.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
score | 2.80 (0.65) | 2.87 (0.91)

13. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Matrix Reasoning
Description: The TestMyBrain Digital Neuropsychology Toolkit Matrix Reasoning task measures abstract reasoning and fluid intelligence by requiring individuals to identify patterns and complete visual matrices.
  In Test my Brain Matrix Reasoning, the participant selects which smaller image completes the pattern in the larger image. This is a test of visual reasoning and general cognitive ability. This test was adapted from the Wechsler Adult Intelligence Scales. Scores go from 2 to 32. Higher scores are better.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Test My Brain Matrix Reasoning.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 28
score | 22.18 (6.52) | 22.58 (6.04)

14. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Serial Reaction Time
Description: The TestMyBrain Digital Neuropsychology Toolkit Serial Reaction Time task measures implicit learning and motor sequence acquisition by assessing response speed to repeating and random stimulus patterns.
  In the TMB Serial Reaction Time task, higher scores in seconds (i.e., longer reaction times) indicate:
  Reduced processing speed Lower motor or attentional efficiency Weaker implicit sequence learning
Time Frame: 4 weeks.
Population: The population included in the analysis was those who completed the Test My Brain Serial Reaction Time.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 29
seconds | 333.24 (60.57) | 384.62 (96.47)

15. Secondary Outcome: Test My Brain Digital Neuropsychology Toolkit - Visual Paired Associates
Description: The TestMyBrain Digital Neuropsychology Toolkit Visual Paired Associates task measures associative memory by requiring individuals to learn and recall visual symbol pairs.
  In this test, the participant memorizes a set of picture pairs. Then, after completing TMB Digit Symbol Matching (90 sec), the participant selects which pictures were paired together. TMB Visual PA is a test of visual episodic memory. In TMB Digit SM, the participant matches as many number/symbol pairs as possible in 90 seconds. This is a test of processing speed. Scores go from 4 to 23. Higher scores are better.
Time Frame: 4 weeks
Population: The population included in the analysis was those who completed the Test My Brain Visual Paired Associates.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 28
score | 16.2 (4.41) | 16.3 (3.93)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from baseline to the last study visit, which included 1 week of baseline measurements, a 4-week exposure period, and 6 study visits, for an estimate of 8 weeks.
Arm/Group | Intervention | Active Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/40
Other Adverse Events (participants affected / at risk) | 0/36 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT06038643/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT06038643/SAP_000.pdf
  • Informed Consent Form (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT06038643/ICF_002.pdf